CLINICAL TRIAL: NCT04579328
Title: Budikadidi: Making Stunting Visible Trial
Brief Title: Impact of Life-size Growth Charts on Understanding of Stunting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tufts University (Other)
Collaborators: Catholic Relief Services (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Merry Fitzpatrick, Senior Researcher, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00000386
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Stunting
Keywords: stunting; height-for-age; behavior change; malnutrition
MeSH Terms: conditions — Growth Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants are assigned to intervention and control groups. At the end of a 3-month intervention, differences in comprehension of messages on stunting will be measured. Additionally, focus groups in the general community will collect information on perceptions of the messages and growth mats.
Who Masked: Outcomes Assessor
Masking Description: enumerators interviewing/testing the participants on their understanding of the messages will not know whether or not the participants have been exposed to the growth mats (intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lessons with Growth Mats (Experimental): Participants, clustered by neighbor groups, will be given lessons on stunting. During the lessons the trainers will use the growth mats to demonstrate their points. In these villages, village-wide events will expose the full community to the messages in combination to the mats.
  Interventions: Behavioral: Exposure to Growth Mats
- Lessons without Mats (No Intervention): Participants, clustered by neighbor groups, will be given lessons on stunting without the aid of the growth mats. In these villages, village-wide events will expose the full community to the messages without the aid of the mats.

INTERVENTIONS:
Behavioral: Exposure to Growth Mats — see arm/group descriptions for description of intervention
  Arms: Lessons with Growth Mats

SUMMARY:
Randomized control trial testing whether exposure to a wall hanging (growth mat) enabling parents to physically compare their children's height against the World Health Organization (WHO) standards for height-for-age in combination with normal messaging on stunting increases parents' understanding and retention of those messages. Both intervention and control groups will receive messages about stunting over a 3-month period, but the intervention group will also be exposed to the growth mats during the 3-month intervention period. Parents in both groups will be tested post intervention on the messages about stunting and scores will be compared.

DETAILED DESCRIPTION:
This study is embedded within a development program implemented by a consortium led by Catholic Relief Services. The program aims to improve child nutrition, in part, through behavior change messaging. Parents have difficulty understanding that stunting is a problem because the high prevalence (57%) means the entire population curve has shifted to the left - a stunted child appears normal when compared to others in the community.

Through previous work, we have designed a wall-hanging like a life-size, color coded growth chart. Using 2 stage sampling, with parents clustered in neighbor groups, neighbor groups have been randomly assigned to intervention or control. Both groups will receive standard lessons on stunting while only the intervention group will have the growth mats incorporated into the lessons. After 3 months of exposure to the lessons, parents will be tested on their understanding of the key lesson points. Scores between groups will be tested for statistical differences. Qualitative focus groups throughout the intervention period will collect information on perception of the message delivery and the utility of the growth mats.

ELIGIBILITY:
Inclusion Criteria:

* membership and regular participation in the selected neighbor groups

Exclusion Criteria:

* extended absence from the village during the intervention period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Understanding of key messages on stunting | after 3 months of exposure to the lessons
  there are multiple key points in the lessons on stunting accompanying the mats. Interviews will test the level of understanding for each key message, combining them into a composite score. Both individual and composite scores will be compared.

SECONDARY OUTCOMES:
Willingness to change behavior | after 3 months of exposure to the lessons
  Interviews will measure self-reported willingness to practice the recommended behaviors to reduce stunting

CONTACTS AND LOCATIONS:
Overall Officials: Merry Fitzpatrick, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw, non-identifiable results from the questions related to understanding of stunting will be available in .xlsx format from the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication of results, estimated October-December 2021
Access Criteria: Researchers seeking to use the data to inform other studies, students conducting class-based research, or practitioners seeking to inform behavior change programs to prevent stunting can receive the raw data and supporting information upon request.